CLINICAL TRIAL: NCT00610766
Title: International PRospective Multicenter Study On RadiaTion Dose Estimates Of Coronary CT AngIOgraphy IN Daily Practice
Acronym: PROTECTION-I
Status: Completed | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: PD Dr. Joerg Hausleiter, Deutsches Herzzentrum
Other Study IDs: GE IDE No. R00107
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Coronary Disease
Keywords: coronary CT angiography; radiation dose estimates
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
Estimation of radiation dose of coronary multislice computed tomography (MSCT) angiography in daily practice in an international, multicenter and vendor-independent trial.

DETAILED DESCRIPTION:
Prospective analysis of cardiac CT angiographies enrolled over 1 month

Collection of 1 axial data set and the "patient dose protocol" (including kV, mAs, CTDI, DLP, etc.) on a CD

Dose estimation in dose/cm with the use of a method proposed by the European Working Group for Guidelines on Quality Criteria in CT.

Assessment of diagnostic, qualitative image quality on a per-vessel basis by the participating study sites and in randomly selected cases by the primary study investigators (approximately 5-10% of patients to "spot check" interobserver variability of image quality assessments)

Assessment of image quality with the use of quantitative parameters including image noise, signal-to-noise and contrast-to-noise ratios

ELIGIBILITY:
Inclusion Criteria:

* assessment of coronary arteries
* acute chest pain or "triple rule out"
* evaluation after PCI (stents)
* evaluation of bypass grafts
* before or after EP study
* cardiac anomalies

Exclusion Criteria:

* pregnancy
* contraindications against contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with indication for cardiac imaging by MSCT
Sampling Method: Non-Probability Sample
Enrollment: 1965 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Radiation dose estimates of coronary MSCT angiography in daily practice | 1 month

SECONDARY OUTCOMES:
Comparison of dose estimates between 16-slice, 64-slice, DSCT and other CT systems | 1 month
Frequency of dose-saving algorithm's use (e.g.: ECG-dose pulsing / Care Dose 4D / 100kv | 1 month
Assessment of potentials for additional dose savings (e.g. entire scan length; the distance between scan start to begin of coronary arteries and distance end of coronary arteries to end of scan) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Hausleiter, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany